CLINICAL TRIAL: NCT00276367
Title: The Impact of Post Discharge One-Time Home Visit: Bridging the Gap Between Hospital and Home.
Status: Withdrawn | Type: Observational
Why Stopped: is involved in NIH study
Sponsor: Maimonides Medical Center (Other)
Other Study IDs: 05/12/02
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: COPD; Coronary Artery Disease; Diabetes Mellitus; Stroke
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Coronary Artery Disease; Diabetes Mellitus; Stroke

SUMMARY:
A single post-hospital discharge home visit by a geriatric nurse practitioner or geriatric fellow can bridge the gap and ease the transition for elderly frail patients returning home after hospital admission. We believe this intervention will reduce medication errors, ensure follow-up discharge plans, decrease re-hospitalization rates, and decrease morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to the ACE unit during the study time frame, age 65 and over, and residing in the community before and after discharge from the hospital. Selected patients will have complex discharge plans including referrals to home care agencies, poly-pharmacy, multiple co-morbidities, history of repeated hospitalizations, and poor social support systems in the community. In addition, eligible patients will have at least one of eight admitting diagnoses, chosen for their high likelihood of requiring post-discharge home care needs. These diagnosis include: CHF, COPD, coronary artery disease, diabetes mellitus, stroke, hip fracture, peripheral vascular disease or cardiac arrhythmia. The GNP or fellow will then request permission from the patient's primary physician to do a one-time post-discharge home visit.

Exclusion Criteria:

Patients discharged to settings other than their homes (i.e. nursing home, sub-acute rehabilitation, etc.)Patients discharged to settings other than their homes (i.e. nursing home, sub-acute rehabilitation, etc.)

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Although IRB approval was received, study was not initiated.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Zagorin, MA, GNP-C, ANP-C, Principal Investigator — Maimonides Medical Center